CLINICAL TRIAL: NCT00883051
Title: A Double Blind Randomized Placebo-Controlled Parallel Group Dose-Ranging Study of Oral COL-144 in the Acute Treatment of Migraine
Brief Title: Dose-ranging Study of Oral COL-144 in Acute Migraine Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: CoLucid Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16892; H8H-CD-LAHO (Other: Eli Lilly and Company); 2008-005010-43 (EudraCT Number); COL MIG-202 (Other: Colucid)
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Results first posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2018-01

CONDITIONS: Migraine Disorders
Keywords: COL-144; acute treatment; migraine
MeSH Terms: conditions — Migraine Disorders | interventions — lasmiditan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 50 mg Lasmiditan (Experimental): 50 mg lasmiditan administered orally (PO)
  Interventions: Drug: Lasmiditan
- 100 mg Lasmiditan (Experimental): 100 mg lasmiditan administered orally (PO)
  Interventions: Drug: Lasmiditan
- 200 mg Lasmiditan (Experimental): 200 mg lasmiditan administered orally (PO)
  Interventions: Drug: Lasmiditan
- 400 mg Lasmiditan (Experimental): 400 mg lasmiditan administered orally (PO)
  Interventions: Drug: Lasmiditan
- Placebo (Placebo Comparator): Placebo administered orally (PO)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lasmiditan — Oral application of one dose of either 50 mg lasmiditan,100 mg lasmiditan, 200 mg lasmiditan, 400 mg lasmiditan or placebo as the first treatment for a new migraine attack providing that any aura symptoms have resolved and the headache is either moderate or severe and has been so for less than 4 hours.
  Other Names: LY573144
  Arms: 100 mg Lasmiditan; 200 mg Lasmiditan; 400 mg Lasmiditan; 50 mg Lasmiditan
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of a range of oral doses of COL-144 in treating migraine headache, in order to select a dose or doses for further evaluation.

DETAILED DESCRIPTION:
Migraine is a common chronic neurological disorder characterized by recurrent disabling episodes of moderate to severe headache accompanied by nausea, vomiting, photophobia, and phonophobia. Acute pharmacologic therapy for migraine aims to terminate the attack or reduce its severity. Analgesics are commonly used or, if these are ineffective, triptans. Since triptans are contraindicated in patients with coronary artery disease, uncontrolled hypertension, and cerebrovascular disease alternative medications are required for patients where simple analgesics do not work. COL-144 has no vasoconstrictor activity at clinically relevant concentrations and might meet this need. COL-144 was effective when given intravenously in a placebo-controlled dose-ranging study. This study investigates which dose of oral COL-144 is effective in the in acute treatment of migraine headache.

ELIGIBILITY:
Inclusion Criteria:

* Patients with migraine with or without aura fulfilling the IHS diagnostic criteria 1.1 and 1.2.1 (2004)
* History of migraine of at least 1 year
* Migraine onset before the age of 50 years
* History of 1 - 8 migraine attacks per month
* Male or female patients aged 18 to 65 years
* Female patients of child-bearing potential must be using a highly effective form of contraception (e.g., combined oral contraceptive, IUD, abstinence, vasectomized partner)
* Able and willing to give written informed consent
* Able and willing to complete a migraine diary card to record details of the attack treated with study medication

Exclusion Criteria:

* History of life threatening or intolerable adverse reaction to any triptan
* Use of prescription migraine prophylactic drugs within 15 days (30 days for flunarizine) prior to Screening Visit and during study participation
* Using herbal preparations (e.g., feverfew, butterbur) for migraine prophylaxis
* Using 5-HT reuptake inhibitors
* Using drugs known to inhibit CYP450 enzymes (see Appendix 2 for details)
* Pregnant or breast-feeding women
* Women of child-bearing potential not using highly effective contraception
* History or evidence of coronary artery disease, ischemic or hemorrhagic stroke, epilepsy or any other condition placing the patient at increased risk of seizures
* History of hypertension (controlled or uncontrolled)
* History of orthostatic hypotension
* Current use of hemodynamically active cardiovascular drugs
* History within the previous 3 years or current evidence of abuse of any drug, prescription or illicit, or alcohol
* Significant renal or hepatic impairment
* Previous participation in this clinical trial
* Participation in any clinical trial of an experimental drug or device in the previous 30 days
* Any medical condition or laboratory test which in the judgment of the investigator makes the patient unsuitable for the study
* Known Hepatitis B or C or HIV infection
* Patients who are employees of the sponsor
* Relatives of, or staff directly reporting to, the investigator
* Patients with known hypersensitivity to COL-144, other 5HT1F receptor agonists or to any excipient of COL-144 drug product
* Patients who were treated with study medication in the COL MIG-201 study (Patients screened but not treated under that protocol are not excluded)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2009-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (38):
- Belgium (6):
  - Montegnée, Liege
  - Hasselt, Limburg
  - Leuven, Vlaams-Brabant
  - Bruges, West-Vlaanderen
  - Brussels
  - Liège
- Finland (7):
  - Helsinki, Etelä-Suomi
  - Hyvinkää, Etelä-Suomi
  - Mikkeli, Itä-Suomen Lääni
  - Pori, Länsi-Suomen
  - Jyväskylä, Länsi-Suomi
  - Tampere, Länsi-Suomi
  - Turku, Länsi-Suomi
- France (6):
  - Nice, Alpes-Maritimes
  - Bordeaux, Gironde
  - Toulouse, Haute-Garonne
  - Lille, Nord
  - Rouen, Seine-Maritime
  - Paris
- Germany (11):
  - Freiburg/Breisgau, Baden-Wurttemberg
  - Göppingen, Baden-Wurttemberg
  - München, Bavaria
  - Wiesbaden, Hesse
  - Erkelenz, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Itzehoe, Schleswig-Holstein
  - Berlin
  - Bremen
  - Hamburg
- Spain (8):
  - Seville, Andalusia
  - Barcelona, Catalonia
  - Santiago de Compostela, Galicia
  - Alcorcón, Madrid
  - Pamplona, Navarre
  - Oviedo, Principality of Asturias
  - Gandia, Valencia
  - Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Blumenfeld A, Tepper SJ, Khanna R, Doty E, Vincent M, Miller SI. Serotonin syndrome in the acute treatment landscape of migraine: the lasmiditan experience. Front Neurol. 2023 Oct 27;14:1291102. doi: 10.3389/fneur.2023.1291102. eCollection 2023. PMID 37965170
- [Derived] Farkkila M, Diener HC, Geraud G, Lainez M, Schoenen J, Harner N, Pilgrim A, Reuter U; COL MIG-202 study group. Efficacy and tolerability of lasmiditan, an oral 5-HT(1F) receptor agonist, for the acute treatment of migraine: a phase 2 randomised, placebo-controlled, parallel-group, dose-ranging study. Lancet Neurol. 2012 May;11(5):405-13. doi: 10.1016/S1474-4422(12)70047-9. Epub 2012 Mar 28. PMID 22459549

RESULTS

PARTICIPANT FLOW:
Groups:
- 50 mg Lasmiditan: 50 mg lasmiditan administered PO within 4 hours of a migraine attack
- 100 mg Lasmiditan: 100 mg lasmiditan administered PO within 4 hours of a migraine attack
- 200 mg Lasmiditan: 200 mg lasmiditan administered PO within 4 hours of a migraine attack
- 400 mg Lasmiditan: 400 mg lasmiditan administered PO within 4 hours of a migraine attack
- Placebo: Placebo administered PO within 4 hours of a migraine attack
Period: Overall Study
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan | 400 mg Lasmiditan | Placebo
Started | 106 | 104 | 100 | 99 | 103
No Study Medication Used | 24 | 22 | 29 | 29 | 17
Received at Least 1 Dose of Study Drug | 82 | 82 | 71 | 70 | 86
Completed | 82 | 82 | 71 | 70 | 85 (One participant was lost to follow up and did not provide adverse event data.)
Not Completed | 24 | 22 | 29 | 29 | 18
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Did not use study medication | 24 | 22 | 29 | 29 | 17

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan | 400 mg Lasmiditan | Placebo | Total
Number analyzed (Participants) | 82 | 82 | 71 | 70 | 86 | 391
Age, Continuous [Median (Full Range); unit: years] | 41 [18 to 65] | 45 [20 to 65] | 41 [18 to 57] | 40 [20 to 60] | 41 [19 to 66] | 41.0 [18.0 to 66.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 68 | 65 | 65 | 75 | 342
  Male | 13 | 14 | 6 | 5 | 11 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 82 | 82 | 71 | 69 | 86 | 390
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 1
  White | 81 | 81 | 70 | 69 | 86 | 387
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants]
  Belgium | 5 | 5 | 6 | 4 | 7 | 27
  Finland | 26 | 26 | 23 | 19 | 30 | 124
  France | 9 | 8 | 5 | 5 | 9 | 36
  Germany | 36 | 34 | 34 | 37 | 32 | 173
  Spain | 6 | 9 | 3 | 5 | 8 | 31

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Headache Response
Description: Headache response is a binary response variable derived from the headache intensities recorded in the participant diary. Headache response is defined as a reduction in headache severity from moderate or severe at baseline to mild or no headache, at two hours after administration of study drug.
Time Frame: 2 hours postdose
Population: All randomized participants who received at least 1 dose of study drug and had a post-baseline evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan | 400 mg Lasmiditan | Placebo
Number analyzed (Participants) | 79 | 81 | 69 | 68 | 81
percentage of participants
  No | 57.0 | 35.8 | 49.3 | 35.3 | 74.1
  Yes | 43.0 | 64.2 | 50.7 | 64.7 | 25.9
Statistical Analysis 1: Comparison: 50 mg Lasmiditan vs 100 mg Lasmiditan vs 200 mg Lasmiditan vs 400 mg Lasmiditan vs Placebo; Test type: Other — A hierarchical test procedure was applied only for analysis of the primary efficacy endpoint; p < 0.0001, Cochran-Armitage test for trend

2. Secondary Outcome: Percentage of Participants Who Are Headache Free (Absence of Headache) After First Dose
Description: The percentage of participants defined as mild, moderate, or severe headache pain becoming none.
Time Frame: 2 hours post dose
Population: All randomized participants who received at least 1 dose of study drug, a 2 hour postdose evaluation and evaluable headache relief data.
Measure: Number; unit: percentage of participants
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan | 400 mg Lasmiditan | Placebo
Number analyzed (Participants) | 79 | 81 | 69 | 68 | 81
percentage of participants | 13.9 | 13.6 | 18.8 | 27.9 | 7.4
Statistical Analysis 1: Comparison: 50 mg Lasmiditan vs 100 mg Lasmiditan vs 200 mg Lasmiditan vs 400 mg Lasmiditan; Test type: Other — A hierarchical test procedure was applied only for analysis of the primary efficacy endpoint; p = 0.0006, Cochran-Armitage test for trend]

3. Secondary Outcome: Percentage of Participants With Headache Recurrence
Description: Participants who received study drug and which became pain free at 2 hours postdose and worsened again upto 24 hours post-dose.
Time Frame: up to 24 hours postdose
Population: Randomized participants who received a dose of study drug, were pain free at 2 hours postdose and had postdose headache severity or symptom assessments.
Measure: Number; unit: percentage of participants
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan | 400 mg Lasmiditan | Placebo
Number analyzed (Participants) | 34 | 52 | 35 | 44 | 21
percentage of participants | 55.9 | 57.7 | 62.9 | 50.0 | 57.1

4. Secondary Outcome: Percentage of Participants With Headache Severity (4 Point Rating Scale)
Description: Headache severity was evaluated by the participant using the International Headache Society (IHS) four point headache severity rating scale (0=no pain, 1=mild pain, 2=moderate pain, and 3=severe pain) with a lower score being less severe and a higher score being more severe.
Time Frame: 2 hours postdose
Population: Randomized participants who received a dose of study drug and had postdose headache severity or symptom assessments.
Measure: Number; unit: percentage of participants
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan | 400 mg Lasmiditan | Placebo
Number analyzed (Participants) | 79 | 80 | 68 | 67 | 81
percentage of participants
  None (0) | 13.9 | 13.6 | 18.8 | 27.9 | 7.4
  Mild(1) | 29.1 | 50.6 | 31.9 | 36.8 | 18.5
  Moderate(2) | 27.8 | 23.5 | 26.1 | 20.6 | 27.2
  Severe(3) | 29.1 | 11.1 | 21.7 | 13.2 | 46.9

5. Secondary Outcome: Percentage of Participants Who Have Symptoms of Nausea
Description: Percentage of participants who have symptoms of nausea two hours post treatment.
Time Frame: 2 hours postdose
Population: Randomized participants who received a dose of study drug and had postdose symptom assessments.
Measure: Number; unit: percentage of participants
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan | 400 mg Lasmiditan | Placebo
Number analyzed (Participants) | 79 | 80 | 68 | 67 | 81
percentage of participants | 31.65 | 25.00 | 35.29 | 26.87 | 40.74

6. Secondary Outcome: Percentage of Participants Who Have Symptoms Phonophobia
Description: Percentage of participants who have symptoms of phonophobia two hours post treatment.
Time Frame: 2 hours postdose
Population: Randomized participants who received a dose of study drug and had postdose symptom assessments.
Measure: Number; unit: percentage of participants
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan | 400 mg Lasmiditan | Placebo
Number analyzed (Participants) | 79 | 80 | 68 | 67 | 81
percentage of participants | 41.77 | 23.75 | 39.71 | 31.34 | 48.15

7. Secondary Outcome: Percentage of Participants Who Have Photophobia
Description: Percentage of participants who have symptoms of photophobia two hours post treatment.
Time Frame: 2 hours postdose
Population: Randomized participants who received a dose of study drug and had postdose symptom assessments.
Measure: Number; unit: percentage of participants
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan | 400 mg Lasmiditan | Placebo
Number analyzed (Participants) | 79 | 80 | 68 | 67 | 81
percentage of participants | 46.84 | 31.25 | 41.18 | 37.31 | 65.43

8. Secondary Outcome: Percentage of Participants With Vomiting
Description: Percentage of participants with vomiting 2 hours post treatment.
Time Frame: 2 hours postdose
Population: Randomized participants who received a dose of study drug and had postdose symptom assessments.
Measure: Number; unit: percentage of participants
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan | 400 mg Lasmiditan | Placebo
Number analyzed (Participants) | 79 | 80 | 68 | 67 | 81
percentage of participants | 5.06 | 0.00 | 7.35 | 4.80 | 11.11

9. Secondary Outcome: Disability (4 Point Scale: Not at All, Mild Interference, Marked Interference, Completely - Needs Bed Rest)
Description: The participant is asked "How much is the migraine interfering with normal activities?" on a 4 point scale 0-Not at all, 1-Mild interference, 2-Marked interference ,3-Completely needs bed rest, with a lower score having lower interference and higher score worse interference.
Time Frame: 2 hours postdose
Population: All randomized participants who received at least 1 dose of study drug and had evaluable data.
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan | 400 mg Lasmiditan | Placebo
Number analyzed (Participants) | 79 | 78 | 66 | 63 | 81
Participants
  Not at all (0) | 13 | 14 | 12 | 10 | 6
  Mild interference (1) | 26 | 33 | 23 | 26 | 23
  Marked interference (2) | 24 | 20 | 17 | 15 | 21
  Completely needs bed rest (3) | 16 | 11 | 14 | 12 | 31

10. Secondary Outcome: Percentage of Participants Who Used Rescue Medication
Description: Rescue medication was permitted after completion of the 2 hour assessment if migraine did not respond (participant was not pain free).
Time Frame: Postdose 2 through 24 hours
Population: Randomized participants who received a dose of study drug and had postdose headache severity or symptom assessments.
Measure: Number; unit: percentage of participants
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan | 400 mg Lasmiditan | Placebo
Number analyzed (Participants) | 79 | 81 | 69 | 69 | 81
percentage of participants | 54.5 | 51.9 | 61.2 | 41.8 | 68.8

11. Secondary Outcome: Number of Participants Reporting a Score on the Patient Global Impression of Improvement (PGI-I)
Description: PGI-I requests participants to mark the box that best describes their cluster headache condition since they started taking the medicine. The options in the displayed boxes are represented on a 7-point scale, with 1 = very much better, 2 = much better, 3 = a little better, 4 = no change, 5 = a little worse, 6 = much worse, and 7 = very much worse, a lower number indicates much better and a higher number indicates worse.
Time Frame: 2 hours postdose
Population: All randomized participants who received at least 1 dose of study drug and had a PGI-I measurement post dose.
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan | 400 mg Lasmiditan | Placebo
Number analyzed (Participants) | 79 | 81 | 69 | 67 | 81
Participants
  Very much better | 3 | 2 | 3 | 4 | 3
  Much better | 15 | 27 | 16 | 19 | 10
  A little better | 28 | 30 | 21 | 22 | 18
  No change | 18 | 11 | 12 | 7 | 27
  A little worse | 7 | 6 | 6 | 9 | 8
  Much worse | 5 | 4 | 3 | 4 | 9
  Very much worse | 3 | 1 | 8 | 2 | 6

12. Secondary Outcome: Actual Time to Headache Relief and Time to Pain Free
Description: The participant answered "Did your migraine pain go away completely (pain free) within 24 hours of dosing" and record the time.
  Actual time to meaningful pain relief and actual time to pain free will be censored at 24 hours if meaningful pain relief or pain free is documented to be greater than 24 hours after dosing and "Did you experience meaningful relief (headache relief) from your migraine within 24 hours after dosing?".
Time Frame: up to 24 hours postdose
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Error); unit: minutes
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan | 400 mg Lasmiditan | Placebo
Number analyzed (Participants) | 79 | 81 | 69 | 68 | 81
minutes
  Pain relief | 650.87 (77.53) | 291.05 (32.24) | 407.16 (52.48) | 218.93 (23.87) | 760.15 (71.19)
  Pain free | 871.27 (72.74) | 767.33 (74.36) | 690.89 (59.67) | 437.12 (36.05) | 1046.47 (77.90)

13. Secondary Outcome: Change From Baseline in Heart Rate
Description: Change from baseline in assessment of vital signs (heart rate).
Time Frame: Baseline through Day 14
Population: Randomized participants who received at least 1 dose of study drug and had evaluable ECG parameters.
Measure: Median (Full Range); unit: beats per minute
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan | 400 mg Lasmiditan | Placebo
Number analyzed (Participants) | 81 | 82 | 71 | 70 | 83
beats per minute | 2.0 [-27.0 to 28.0] | 3.0 [-16.0 to 24.0] | 1.0 [-18.0 to 28.0] | 2.0 [-21.0 to 28.0] | 1.0 [-66.0 to 18.0]

14. Secondary Outcome: Change From Baseline in Systolic Blood Pressure
Description: Change from baseline in vital signs (systolic blood pressure).
Time Frame: Baseline through Day 14
Population: All randomized participants who received at least 1 dose of study drug and had evaluable blood pressure.
Measure: Median (Full Range); unit: millimeters of mercury
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan | 400 mg Lasmiditan | Placebo
Number analyzed (Participants) | 82 | 82 | 70 | 70 | 83
millimeters of mercury | 1.0 [-30.0 to 29.0] | 0.0 [-25.0 to 42.0] | -1.5 [-23.0 to 35.0] | -0.5 [-35.0 to 36.0] | -0.0 [-30.0 to 35.0]

15. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure
Description: Change from baseline in vital signs (diastolic blood pressure).
Time Frame: Baseline through Day 14
Population: Randomized participants who received at least 1 dose of study drug and had evaluable blood pressure.
Measure: Median (Full Range); unit: millimeters of mercury
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan | 400 mg Lasmiditan | Placebo
Number analyzed (Participants) | 82 | 82 | 70 | 70 | 83
millimeters of mercury | 0.0 [-14.0 to 21.0] | 0.0 [-20.0 to 25.0] | 0.0 [-22.0 to 15.0] | 0.0 [-20.0 to 20.0] | 0.0 [-20.0 to 21.0]

16. Secondary Outcome: Percentage of Participants With Change From Baseline in Physical Examination Parameters
Description: Participants were evaluated for skin, head, ear, nose and throat, cardiovascular and musculoskeletal changes from a normal screening to an abnormal screening. Changes in the physical examination noted as non-serious AEs or SAEs, regardless of causality, are located in the Reported Adverse Events section.
Time Frame: Baseline through Day 14
Population: All randomized participants who received at last 1 dose of study drug and had a physical examination.
Measure: Number; unit: percentage of participants
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan | 400 mg Lasmiditan | Placebo
Number analyzed (Participants) | 82 | 82 | 71 | 70 | 86
percentage of participants
  Skin | 1.2 | 2.4 | 1.4 | 0 | 0
  Head, ears, nose, throat | 0 | 0 | 0 | 1.4 | 0
  Musculoskeletal | 0 | 1.2 | 0 | 0 | 3.5

17. Secondary Outcome: Change From Baseline in Hematology Tests
Description: Hematology tests, including a complete blood count (CBC) measured red blood cells, white blood cells, hemoglobin, neutrophils and platelets.
Time Frame: Baseline through Day 14
Population: All randomized participants who received at least 1 dose of study drug and had evaluable blood parameters.
Measure: Mean (Standard Error); unit: million cells per liter
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan | 400 mg Lasmiditan | Placebo
Number analyzed (Participants) | 82 | 82 | 71 | 70 | 84
million cells per liter
  Hemoglobin | 0.0 (0.4) | 0.0 (0.4) | 0.1 (0.4) | 0.0 (0.4) | 0.0 (0.4)
  Red blood cells | 0.0 (0.2) | 0.0 (0.2) | 0.0 (0.2) | 0.0 (0.2) | 0.0 (0.2)
  White blood cells | -0.1 (1.3) | 0.3 (1.4) | -0.3 (1.6) | -0.4 (1.7) | -0.2 (1.6)
  Neutrophils | -3.2 (9.3) | -0.3 (7.9) | -2.8 (14.7) | -3.2 (14.7) | -3.9 (9.9)
  Platelets | -2.3 (35.2) | -0.5 (25.9) | 4.6 (48.4) | 2.9 (34.7) | 1.7 (34.7)

18. Secondary Outcome: Number of Serious Adverse Events
Description: A summary of non-serious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: up to 8 weeks
Population: All randomized participants who received at least 1 dose of study drug excluding one participant who was lost to follow-up and did not report adverse events.
Measure: Number; unit: adverse events
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan | 400 mg Lasmiditan | Placebo
Number analyzed (Participants) | 82 | 82 | 71 | 70 | 85
adverse events | 0 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 8 weeks
Description: All randomized participants who received at least 1 dose of study drug excluding one participant from the placebo group who did not report adverse events and was lost to follow up.
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan | 400 mg Lasmiditan | Placebo
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/82 | 0/71 | 0/70 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/82 | 1/71 | 0/70 | 0/85
Other Adverse Events (participants affected / at risk) | 53/82 | 59/82 | 60/71 | 59/70 | 19/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50 mg Lasmiditan (N=82) | 100 mg Lasmiditan (N=82) | 200 mg Lasmiditan (N=71) | 400 mg Lasmiditan (N=70) | Placebo (N=85)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50 mg Lasmiditan (N=82) | 100 mg Lasmiditan (N=82) | 200 mg Lasmiditan (N=71) | 400 mg Lasmiditan (N=70) | Placebo (N=85)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 8 (8) | 12 (12) | 12 (12) | 16 (16) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Halo vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 8 (8) | 2 (2) | 5 (6) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 3 (3) | 7 (7) | 2 (2) | 4 (4) | 0 (0)
Chest discomfort (General disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Discomfort (General disorders) | 2 (2) | 2 (2) | 4 (4) | 4 (4) | 2 (2)
Fatigue (General disorders) | 10 (11) | 17 (17) | 15 (15) | 16 (16) | 2 (2)
Feeling abnormal (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 3 (3) | 4 (4) | 2 (2) | 1 (1) | 1 (1)
Feeling hot (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Feeling of body temperature change (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling of relaxation (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Malaise (General disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sensation of blood flow (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5) | 4 (4) | 3 (3) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Coordination abnormal (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1) | 3 (4) | 1 (1) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 19 (21) | 21 (22) | 26 (26) | 26 (27) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fine motor delay (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 3 (4) | 5 (5) | 4 (5) | 1 (1)
Hypotonia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 9 (9) | 12 (16) | 14 (14) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sedation (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Slow response to stimuli (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 8 (8) | 10 (11) | 8 (9) | 8 (8) | 2 (3)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Derealisation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Euphoric mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fear (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Illusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
One participant from the placebo group did not report adverse events and was lost to follow up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days